CLINICAL TRIAL: NCT03157570
Title: Effects of Home Exercise Intervention on Bone Density, Muscle Functions, Quality of Life, and Curve Progression in Girls With Adolescent Idiopathic Scoliosis
Brief Title: Effects of Home Exercise Intervention on Bone Density, Muscle Functions, QoL, and Curve Progression in Girls With AIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Man Shan Elisa Tam, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AISE_20170407
Record Dates: First submitted 2017-05-08; First posted 2017-05-17 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Adolescent Idiopathic Scoliosis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention group (Experimental): The exercise group will participate in a 6-month home exercise along with demonstration videos. The exercise training program is an online 7-minute high-intensity interval training (HIIT) exercise through the integrated application of an exercise provision website and mobile Apps. The program will comprise of a broad range of exercises, applied at varying speeds and directions in order to increase heart rate, and to load a variety of muscle groups and skeletal regions in the upper and lower body. The exercise will be performed 5 days per week with the remaining 2 days as rest days.
  Interventions: Behavioral: Exercise
- Control group (No Intervention): The control group have no intervention and receives only standard care.

INTERVENTIONS:
Behavioral: Exercise — 7-min High Intensity Interval Training with 12 different exercises (each exercise 30 seconds continuously with 10 seconds rest interval)
  Arms: Exercise intervention group

SUMMARY:
Studies with exercise intervention aimed to improve the bone health and muscle functions in patients with AIS were lacking. Evidence suggested that low bone mass and low muscle mass were associated with curve severity and occurrence of AIS. Weight-bearing exercise that aimed to improve musculoskeletal and metabolic health could enhance bone health and muscle mass, and could provide a feasible alternative conservative treatment to prevent curve progression as well as the quality of life in AIS girls. This is a pilot feasibility study for future large randomized controlled trial (RCT) aiming at determining the effects of home based exercise program on improving bone mineral density (BMD), muscle mass and functions, quality of life (QoL), and prevent curve progression in skeletally immature girls with adolescent idiopathic scoliosis (AIS).

ELIGIBILITY:
Inclusion Criteria:

* Cobb Angle greater or equal to 15°
* Newly diagnosed at the Scoliosis Clinic without prior treatment
* Cleared for physical activity by doctor

Exclusion Criteria:

* Scoliosis with any known etiology such as congenital scoliosis, neuromuscular scoliosis, scoliosis of metabolic etiology, scoliosis with skeletal dysplasia, or
* Known endocrine and connective tissue abnormalities, or
* Known heart condition or other diseases that could affect the safety of exercise
* Eating disorders or GI malabsorption disorders or
* Currently taking medication that affects bone or muscle metabolism

Ages: 11 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Change in BMD after completion of exercise | Baseline and 6 months
  Areal BMD (g/cm2) of non-dominant femoral neck and greater trochanter, and whole body BMD will be measured by DXA (Horizon, Hologic Inc., USA). Standardized scanning procedure provided by the manufacturer will be followed to ensure unified and comparable measurement. Quality assurance is performed by daily calibration against the standard phantoms provided by the manufacturer, with a precision error of 1.9% for BMD value for patient scan and <1.0% for whole body phantom scan.
Change in Muscle mass after completion of exercise | Baseline and 6 months
  Muscle mass will be measurement by whole body less head (WBLH) scan with DXA (Horizon, Hologic Inc., USA). DXA is the current golden standard to the measurement of body composition. Standardized scanning procedure provided by the manufacturer will be followed to ensure unified and comparable measurement.
Change in Anthropometric measurements after completion of exercise | Baseline and 6 months
  Body height, weight, sitting height, and arm span will be measured with standard stadiometry techniques.
Change in BMC after completion of exercise | Baseline and 6 months
  BMC (g/cm) of non-dominant femoral neck and greater trochanter, and whole body BMC will be measured by DXA (Horizon, Hologic Inc., USA). Standardized scanning procedure provided by the manufacturer will be followed to ensure unified and comparable measurement.

SECONDARY OUTCOMES:
Change in clinical features after completion of exercise | Baseline and 6 months
  A long standard standing postero-anterior (PA) whole spine radiograph will be used for grading curve severity in terms of Cobb angle according to the standard Cobb method. Risser sign, curve level and apex, and curve type will be recorded as in any standard assessment of scoliosis patients.
Change in clinical features 1 year after completion of exercise | Baseline and 18 months
  A long standard standing postero-anterior (PA) whole spine radiograph will be used for grading curve severity in terms of Cobb angle according to the standard Cobb method. Risser sign, curve level and apex, and curve type will be recorded as in any standard assessment of scoliosis patients.
Change in muscle strength after completion of exercise | Baseline and 6 months
  Legs, back, abdominal, and handgrip muscle strength will be assessed with dynamometer. The tests will be performed 3 times with 1 familiarization effort and 2 maximal effort, and the highest scores will be used for analysis.
Change in muscle strength 1 year after completion of exercise | Baseline and 18 months
  Legs, back, abdominal, and handgrip muscle strength will be assessed with dynamometer. The tests will be performed 3 times with 1 familiarization effort and 2 maximal effort, and the highest scores will be used for analysis.
Change in muscle endurance after completion of exercise | Baseline and 6 months
  Isometric squat test, Biering-Sorensen test, and isometric curl-up test will be used to assess the quadriceps, back and abdominal muscle endurance. The time (seconds) in which the subject maintained the position is recorded.
Change in muscle endurance 1 year after completion of exercise | Baseline and 18 months
  Isometric squat test, Biering-Sorensen test, and isometric curl-up test will be used to assess the quadriceps, back and abdominal muscle endurance. The time (seconds) in which the subject maintained the position is recorded.
Change in aerobic fitness after completion of exercise | Baseline and 6 months
  Aerobic fitness (estimated VO2max) of the subjects will be measured using sing-stage cycle ergometer sub-maximal test. Participants will be asked to sit on a cycle ergometer with 3-5 min warm up cycling at 150 kgm/min (25 Watt) workload, then workload will increase to 450-600 kgm/min (75-100 Watt) for another 6 minutes, in order to stimulate a submaximal exercise heart rate between 125-170 bpm. Estimated VO2max is then computed from the Astrand formula: VO2max = (workload x 2 + 300) * (200 - 73) / (exercise heart rate - 73)". Safety guidelines and procedures recommended by the ACSM will be followed.
Change in aerobic fitness 1 year after completion of exercise | Baseline and 18 months
  Aerobic fitness (estimated VO2max) of the subjects will be measured using sing-stage cycle ergometer sub-maximal test. Participants will be asked to sit on a cycle ergometer with 3-5 min warm up cycling at 150 kgm/min (25 Watt) workload, then workload will increase to 450-600 kgm/min (75-100 Watt) for another 6 minutes, in order to stimulate a submaximal exercise heart rate between 125-170 bpm. Estimated VO2max is then computed from the Astrand formula: VO2max = (workload x 2 + 300) * (200 - 73) / (exercise heart rate - 73)". Safety guidelines and procedures recommended by the ACSM will be followed.
Change in quality of life after completion of exercise | Baseline and 6 months
  The Quality of Life of the subjects will be assessed with the official Chinese version of Scoliosis Research Society-22 (SRS-22r) Questionnaire. SRS-22r is an internationally validated questionnaire that contains 22 questions organized in 5 domains covering different aspects of the quality of life of patients with scoliosis: function/activity, pain, self-image, mental health (5 items each), and satisfaction with treatment (2 items).
Change in quality of life 1 year after completion of exercise | Baseline and 18 months
  The Quality of Life of the subjects will be assessed with the official Chinese version of Scoliosis Research Society-22 (SRS-22r) Questionnaire. SRS-22r is an internationally validated questionnaire that contains 22 questions organized in 5 domains covering different aspects of the quality of life of patients with scoliosis: function/activity, pain, self-image, mental health (5 items each), and satisfaction with treatment (2 items).
Change in BMD 1 year after completion of exercise | Baseline and 18 months
  Areal BMD (g/cm2) of non-dominant femoral neck and greater trochanter, and whole body BMD will be measured by DXA (Horizon, Hologic Inc., USA). Standardized scanning procedure provided by the manufacturer will be followed to ensure unified and comparable measurement. Quality assurance is performed by daily calibration against the standard phantoms provided by the manufacturer, with a precision error of 1.9% for BMD value for patient scan and <1.0% for whole body phantom scan.
Change in BMC 1 year after completion of exercise | Baseline and 18 months
  BMC (g/cm) of non-dominant femoral neck and greater trochanter, and whole body BMC will be measured by DXA (Horizon, Hologic Inc., USA). Standardized scanning procedure provided by the manufacturer will be followed to ensure unified and comparable measurement.
Change in muscle mass 1 year after completion of exercise | Baseline and 18 months
  Muscle mass will be measurement by whole body less head (WBLH) scan with DXA (Horizon, Hologic Inc., USA). DXA is the current golden standard to the measurement of body composition. Standardized scanning procedure provided by the manufacturer will be followed to ensure unified and comparable measurement.
Change in Anthropometric measurements 1 year after completion of exercise | Baseline and 18 months
  Body height, weight, sitting height, and arm span will be measured with standard stadiometry techniques.

OTHER OUTCOMES:
Recruitment rate | 6 months
  The recruitment rate will be calculated based on the number of eligible subjects invited to the study and the number of eligible subjects agreed to participate.
Dropout rate | 6 months
  The dropout rates for the intervention and control groups will be calculated based on the number of recruited subjects in each group and the number of recruited subjects who failed to complete the 6-month exercise and complete all follow-up.
Dietary intake measures | Baseline, 6 months 18 months
  Evaluation of habitual dietary intake will be based on retrospective means of assessment. A modified Food Frequency Questionnaire (FFQ) based on data obtained in the Hong Kong Adult Dietary Survey in 1995 will be used. The FFQ had been validated with the basal metabolic rate calculation and the 24-hour sodium/creatinine and potassium/creatinine analysis. Subjects will be asked about their usual frequency and consumption in the past twelve months from the food list. Standard portion size will be listed and a food photo album is provided to assist assessment. Any use of supplements will also be recorded. Daily nutrient intake is calculated by the Food Processor Nutrition analysis and Fitness software version 8.0 (Esha Research, Salem, USA), with addition of composition of some local foods based on food composition table from China.
Physical activity measures | Baseline, 6 months 18 months
  Physical activity level will be assessed with a physical activity bracelet and questionnaire. The subjects will be asked to wear the physical activity bracelet every day during the study period, thus provide an objective assessment of the physical activity of the wearer. Physical activity level of the subjects will also be assessed with the modified Baecke questionnaire adapted from Pols et al.
Maturity assessment | Baseline, 6 months 18 months
  Sexual maturity level including the breast development, onset of menarche, pubic hair distribution will be graded with standard Tanners Scale using the established and validated protocols.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong